CLINICAL TRIAL: NCT05246462
Title: The Effect of Logotherapy on Traumatic Stress Symptom, Post-Traumatic Growth, Finding Meaning in Life, and Spiritual Well-Being in Gynecological Cancer Patients: A Randomized Control Study
Brief Title: The Effect of Logotherapy on Mental Health in Gynecological Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ruveyde AYDIN, Akdeniz University Health Sciences Institute, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/48); Ruveyde AYDIN (Registry Identifier: Ruveyde AYDIN)
Record Dates: First submitted 2022-01-12; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Cancer of Ovary; Endometrium Cancer; Cervix Cancer
Keywords: gynecological cancers; post-traumatic growth; the meaning of life; nursing; logotherapy
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms | interventions — Logotherapy

STUDY DESIGN:
Intervention Model Description: This study was conducted between 25 March-15 December 2019 as a single-blind randomized controlled trial.
Who Masked: Participant
Masking Description: Participants were blinded to treatment allocation. The investigator delivered the intervention and, therefore, could not be blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Gynecological cancer patients in a chemotherapy unit in Trabzon were recruited in the study. Inclusion criteria for the study were volunteering to take part in the study, being able to read and write in Turkish, being 18 years of age or older, having been diagnosed with gynecological cancer, knowing that s/he had been diagnosed with cancer, having received at least one chemotherapy treatment and having cancer stage 2 or 3. Exclusion criteria in the study were having a verbal communication disability, having been diagnosed with psychotic and neurological disorders, having received, or receiving psychotherapy, living outside the city center of Trabzon, and receiving treatment at intervals longer than 21 days. The experimental group received 7 sessions of logotherapy interviews.
  Interventions: Other: Logotherapy
- Control group (No Intervention): Gynecological cancer patients in a chemotherapy unit in Trabzon were recruited in the study. Inclusion criteria for the study were volunteering to take part in the study, being able to read and write in Turkish, being 18 years of age or older, having been diagnosed with gynecological cancer, knowing that s/he had been diagnosed with cancer, having received at least one chemotherapy treatment and having cancer stage 2 or 3. Exclusion criteria in the study were having a verbal communication disability, having been diagnosed with psychotic and neurological disorders, having received, or receiving psychotherapy, living outside the city center of Trabzon, and receiving treatment at intervals longer than 21 days. The control group received standard nursing care.

INTERVENTIONS:
Other: Logotherapy — In this study, the experimental group received seven-session logotherapy-based interviews on making sense of life, while the control group received only routine nursing care. In this study, Personal Meaning Oriented Psychotherapy (PMOP) was used to structure interviews on making sense of life based on Logotherapy and enhance the sense of meaning in cancer patients, share their concerns, experiences, and feelings about diagnosis-treatment, have their difficulties defined, maintain, and develop their sense of purpose and responsibility.
  Arms: Experimental group

SUMMARY:
Gynecological cancers negatively affect women's sexuality, fertility, body image, and self-perception, resulting in deterioration in their psychological health. The aim of this study is to examine the effects of logotherapy on traumatic stress symptoms, post-traumatic growth, finding meaning in life, and spiritual well-being in gynecological cancer patients. No research has yet been found that examines logotherapy's symptoms of post-traumatic stress, post-traumatic growth, the meaning of life, and the spiritual well-being of gynecological cancer patients. The study was conducted in a single-blind randomized controlled trial with 68 women with gynecological cancer. The study is registered at ClinicalTrials.gov NCT… While logotherapy interviews including seven sessions were made in the experimental group, only routine nursing care was given to the control group. The data were collected using the Personal Information Form (PIF), the Traumatic Stress Symptom Scale (TSSS), the Post-Traumatic Growth Inventory (PTGI), the Meaning in Life Questionnaire (MLQ), and the Spiritual Well-Being Scale (SWBS). To analyze the data, descriptive statistics and parametric-nonparametric tests were used in the analysis of the data.

DETAILED DESCRIPTION:
Cancer exposes the individual to challenging situations like lack of knowledge about the treatment process, low/absence of social support, economic difficulties, fear of losing health, changes in roles in society and family, and fear of death. In addition to these situations encountered in all types of cancer, gynecological cancers also negatively affect women's sexuality, fertility, menopause symptoms, and self-perception, leading to the deterioration of their psychological health. The absence of supportive care against these cancer-induced adverse conditions causes stress, anxiety, depression, post-traumatic stress disorder (PTSD), and existential emptiness in patients.

Studies conducted with women with gynecological cancer have shown that the frequency of women experiencing PTSD varies between 9.25% and 70%, and women experience at least two of the symptoms of PTSD. Cancer patients report that they feel lonely, they can hardly control their anger, they are disappointed, they feel unhappy and meaningless. Studies focusing on the experiences of cancer patients have revealed that nearly half of the patients experience meaninglessness and hopelessness. Therefore, it is the primary responsibility of health professionals/nurses to accompany and contribute to the journey of cancer patients to find meaning.

Research Hypotheses

1. The total mean TSSS score of the women in the experimental group who participated in the logotherapy interviews was lower than that of the women in the control group (H1).
2. The total mean PTGI score of the women in the experimental group who participated in the logotherapy interviews was higher than that of the women in the control group (H1).
3. The total mean MLQ score of the women in the experimental group who participated in the logotherapy interviews was higher than that of the women in the control group (H1).
4. The total mean SWBS score of the women in the experimental group who participated in the logotherapy interviews was higher than that of the women in the control group (H1).

ELIGIBILITY:
Inclusion Criteria:

* Gynecological cancer patients in a chemotherapy unit in Trabzon were recruited in the study
* Inclusion criteria for the study were volunteering to take part in the study
* Being able to read and write in Turkish
* Being 18 years of age or older
* Having been diagnosed with gynecological cancer
* Knowing that s/he had been diagnosed with cancer
* Having received at least one chemotherapy treatment and having cancer stage 2 or 3.

Exclusion Criteria:

* Exclusion criteria in the study were having a verbal communication disability
* Having been diagnosed with psychotic and neurological disorders
* Having received, or receiving psychotherapy, living outside the city center of Trabzon
* Receiving treatment at intervals longer than 21 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Traumatic Stress Symptoms Scale (TSSS) | It varies between 7-14 weeks.
  TSSS is a 4-point Likert scale (0=not disturbing at all, 3=very disturbing) and consists of 23 items. The scale includes two sub-dimensions: post-traumatic stress disorder (PTSD) and depression. The lowest score to be obtained from the scale is 0 and the highest score is 69. The total Cronbach's alpha of the scale is 0.94
Post-Traumatic Growth Inventory (PTGI) | It varies between 7-14 weeks.
  The scale consists of 23 items and 5 factors such as spiritual and existential change, change in perception of life and selfness, relating to others, new possibilities, and personal strength. Scoring of the Likert-type scale varies between 0 (never experienced) and 5 (experienced a lot). The lowest score to be taken from the scale is 0, and the highest score is 115. The total Cronbach's alpha of the scale is 0.93.
Meaning in Life Questionnaire (MLQ) | It varies between 7-14 weeks.
  The scale consists of 10 items in total on the scale, and the 9th item is reverse coded. The scale consists of two factors: the presence of meaning and the search for meaning. The scale is scored as a 7-point Likert type (1: not true at all; 7: absolutely true). The lowest and the highest score to be obtained from the scale are 10 and the highest score is 70. The overall Cronbach alpha of the scale is 0.86.
Spiritual Well-Being Scale (SWBS) | It varies between 7-14 weeks.
  The scale consists of 29 items and three sub-dimensions: transcendence, nature harmony, and anomie. The scale is a 5-point Likert type (1: not suitable for me at all, 5: completely suitable for me). The lowest and highest scores to be obtained from the scale are 29 and 145. The total Cronbach alpha of the scale is 0.88.

CONTACTS AND LOCATIONS:
Overall Officials: Akdeniz University Health Sciences Institute, Principal Investigator — Akdeniz University Health Sciences Institute
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (+90), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aydin R, Kabukcuoglu K. The effect of logotherapy-based, nurse-guided meaning attribution conversations on women diagnosed with gynecologic cancer: A Turkish pilot study. Women Health. 2023 Sep 14;63(8):599-614. doi: 10.1080/03630242.2023.2249123. Epub 2023 Aug 29. PMID 37642347